CLINICAL TRIAL: NCT02355379
Title: Randomised Phase III Study Evaluating Adjuvant Chemotherapy After Resection of Stage III Colonic Adenocarcinoma in Patients of 70 and Over Intergroup Trial: Ffcd, Gercor, Gerico, Unicancer-gi
Brief Title: Randomised Study Evaluating Adjuvant Chemotherapy After Resection of Stage III Colonic Adenocarcinoma in Patients of 70 and Over
Acronym: ADAGE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE34-ADAGE
Record Dates: First submitted 2015-01-26; First posted 2015-02-04 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Colonic Adenocarcinoma
Keywords: Adjuvant chemotherapy in colonic adenocarcinoma in elderly
MeSH Terms: conditions — Colonic Neoplasms | interventions — XELOX; Observation; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GROUP1 -ARM A (Experimental): LV5FU2 or capecitabine
  Interventions: Drug: LV5FU2 or capectitabine
- GROUP1-ARMB (Experimental): FOLFOX4 or XELOX
  Interventions: Drug: FOLFOX4 or XELOX
- GROUP2- ARM C (Experimental): Observation
  Interventions: Other: Observation
- GROUP2-ARM D (Experimental): LV5FU2 or capecitabine
  Interventions: Drug: LV5FU2 or capecitabine

INTERVENTIONS:
Drug: LV5FU2 or capectitabine
  Arms: GROUP1 -ARM A
Drug: FOLFOX4 or XELOX
  Arms: GROUP1-ARMB
Other: Observation
  Arms: GROUP2- ARM C
Drug: LV5FU2 or capecitabine
  Arms: GROUP2-ARM D

SUMMARY:
Colorectal cancer occurs mainly in elderly patients. Recent estimation showed that in France more than 50% of the patients diagnosed with a colorectal cancer are 70 years old or more. Adjuvant chemotherapy has demonstrated a benefit on disease-free survival and overall survival after a stage III colon cancer resection. Nevertheless adjuvant chemotherapy is poorly used in elderly patients. Prognostic improvement with chemotherapy based on 5FU is suggested by a post-hoc analysis of randomized prospective clinical trial. But elderly patients in this study were highly selected and patients older than 80 represented only 0.7% of the total population. Thus, there is still a concern about the benefit of adjuvant 5FU-based chemotherapy in very elderly unselected patients.

The recommended treatment for stage III adjuvant chemotherapy is a combination of fuoropyrimidine and oxaliplatin. Nevertheless oxaliplatin did not demonstrated survival advantage in elderly patients.

Altogether there are still two matters of debate:

* First, is there a benefit of fluoropyrimidine-based adjuvant chemotherapy for unfit elderly patients?
* Second, is there a benefit of oxaliplatin-based adjuvant chemotherapy for fit elderly patients? The aim of this randomized phase III study is to evaluate the benefit for disease-free survival of adjuvant chemotherapy in elderly patient and which chemotherapy.

The elderly patient population will be dichotomized into two groups according to physician's choice after a multidisciplinary evaluation involving a geriatrician, with two different randomization assignments. The patients with an expected life-expectancy below 4 years according Lee score are excluded of this study.

Some biological tumour abnormalities are more frequently observed in elderly (i.e. mismatch repair deficiency), therefore an evaluation of specific biological prognostic factors is needed in elderly population.

DETAILED DESCRIPTION:
Colorectal cancer occurs mainly in elderly patients. Recent estimation showed that in France more than 50% of the patients diagnosed with a colorectal cancer are 70 years old or more. Adjuvant chemotherapy has demonstrated a benefit on disease-free survival and overall survival after a stage III colon cancer resection. Nevertheless adjuvant chemotherapy is poorly used in elderly patients. Prognostic improvement with chemotherapy based on 5FU is suggested by a post-hoc analysis of randomized prospective clinical trial. But elderly patients in this study were highly selected and patients older than 80 represented only 0.7% of the total population. Thus, there is still a concern about the benefit of adjuvant 5FU-based chemotherapy in very elderly unselected patients.

The recommended treatment for stage III adjuvant chemotherapy is a combination of fuoropyrimidine and oxaliplatin. Nevertheless oxaliplatin did not demonstrated survival advantage in elderly patients.

Altogether there are still two matters of debate:

* First, is there a benefit of fluoropyrimidine-based adjuvant chemotherapy for unfit elderly patients?
* Second, is there a benefit of oxaliplatin-based adjuvant chemotherapy for fit elderly patients? The aim of this randomized phase III study is to evaluate the benefit for disease-free survival of adjuvant chemotherapy in elderly patient and which chemotherapy.

The elderly patient population will be dichotomized into two groups according to physician's choice after a multidisciplinary evaluation involving a geriatrician, with two different randomization assignments. The patients with an expected life-expectancy below 4 years according Lee score are excluded of this study.

Some biological tumour abnormalities are more frequently observed in elderly (i.e. mismatch repair deficiency), therefore an evaluation of specific biological prognostic factors is needed in elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Patient considered able to receive chemotherapy
* Lee score detailed faxed to CRGA
* Stage III colon adenocarcinoma
* R0 resection of the primary tumor
* Start of the potential adjuvant chemotherapy within 12 weeks after surgery
* No prior chemotherapy for colon cancer
* Geriatric Self-administered questionnaire completed faxed to CRGA
* Geriatric Questionnaire completed by the team faxed to CRGA
* Effective contraception for men patients throughout treatment and for at least 6 months after discontinuation of oxaliplatin
* Consent signed

Exclusion Criteria:

* Other progressive disease (cancer uncontrolled for less than 2 years)
* Rectal Cancer (located less than 15 cm from the anal verge endoscopy or sub-peritoneal)
* ANC <2000 / mm3 for group 1 and ANC <1500 / mm3 for group 2 and platelets <100,000 / mm3 or hemoglobin <9 g / dL
* Neuropathy for patients in group 1
* Known deficit of dihydropyrimidine dehydrogenase (DPD)
* Patients with severe hepatic insufficiency
* Any contrindication to the drugs used in the study
* Inability to submit to medical follow-up for geographical, social or psychological reasons.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 774 (Estimated)
Dates: Start 2015-01; Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The 3-year disease-free survival | 3 years after last patient in

SECONDARY OUTCOMES:
Overal survival | 5 years after last patient in
Observed toxicities, graded according to NCI-CTC v4 | 3 years after last patient in

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aparicio, Pr, Principal Investigator — FFCD member
Locations (137):
- France (137):
  - CHU de Fort de France, Fort de France, Guadeloupe
  - CH d'Abbeville, Abbeville
  - CROMG, Agen
  - Centre hospitalier du Pays d'Aix, Aix-en-Provence
  - Centre hospitalier d'Albi, Albi
  - Clinique Claude Bernard, Albi
  - Centre Oncogard, Alès
  - Hôpital Sud, Amiens
  - ICO Site Paul Papin, Angers
  - CHU d'Angers, Angers
  - HOP Privé, Annemasse
  - CH Victor Dupouy, Argenteuil
  - Hôpital Les Bonnettes, Arras
  - Hôpital Privé Bonnettes, Arras
  - Centre Hospitalier Ardèche Méridionale, Aubenas
  - CH D'Auxerre, Auxerre
  - Hôpital Henri Duffaut, Avignon
  - Institut Sainte Catherine, Avignon
  - Hôpital de Bayeux, Bayeux
  - Centre d'Oncologie et de Radiothérapie du Pays-Basque, Bayonne
  - CH Côte Basque, Bayonne
  - CH de Beauvais, Beauvais
  - CH de Béziers, Béziers
  - CH de Blois, Blois
  - CHU Avicenne, Bobigny
  - Polyclinique Bordeaux Nord, Bordeaux
  - Hôpital Duchenne, Boulogne-sur-Mer
  - Hôpital Pierre Oudot, Bourgoin
  - Clinique Pasteur Saint Esprit, Brest
  - CHU Côte de Nacre, Caen
  - CH, Cahors
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - CH William Morey, Chalon-sur-Saône
  - Hôpital Privé Sainte Marie, Chalon-sur-Saône
  - Centre Hospitalier Métropole Savoie, Chambéry
  - Centre Hospitalier Général, Châlons-en-Champagne
  - Centre Hospitalier Public du Cotentin, Cherbourg
  - CH, Cherbourg
  - CHU Estaing, Clermont-Ferrand
  - Hopitaux Civils de Colmar, Colmar
  - Centre Hospitalier, Compiègne
  - CH, Contamine-sur-Arve
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Clinique des Cèdres, Cornebarrieu
  - Centre Hospitalier de Dax, Dax
  - Service de médecine, Digne-les-Bains
  - Institut de Cancérologie de Bourgogne - GRRECC, Dijon
  - Centre Goerges François Leclerc, Dijon
  - Hôpital François Mitterand, Dijon
  - CHI Elbeuf-Louviers-Val de Reuil, Elbeuf
  - Centre médical des Forcilles, Férolles-Attilly
  - CH, Flers
  - CHI de Fréjus Saint-Raphaël, Fréjus
  - Centre Hospitalier, Gap
  - Centre Hospitalier, Gonesse
  - CH, Gonesse
  - CHU de Grenoble - Hôpital A. Michallon, Grenoble
  - CH Marne La Vallée-Jossigny, Jossigny
  - CHD Vendée, La Roche-sur-Yon
  - Groupe Hospitalier de la Rochelle Ré-Aunis, La Rochelle
  - CH, Le Coudray
  - CH du Mans, Le Mans
  - Centre Oscar Lambret, Lille
  - CHRU Hôpital Claude Huriez 4eme EST, Lille
  - Clinique François Chénieux, Limoges
  - CHU Dupuytren, Limoges
  - CH, Longjumeau
  - CHBS - Hôpital du Scorff, Lorient
  - Clinique Mutualiste Eugène André, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Clinique de la Sauvegarde, Lyon
  - CHU de Lyon - Croix Rousse, Lyon
  - CH ST Joseph-ST Luc, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Européen Marseille, Marseille
  - CHU La Timone, Marseille
  - Hopital Nord, Marseille
  - Centre Radiologie, Mâcon
  - CH de Meaux, Meaux
  - Hôpital Layne, Mont-de-Marsan
  - Centre Hospitalier, Montélimar
  - Hôpital Monod, Montivilliers
  - Centre Hospitalier, Morlaix
  - Centre Azuréen de Cancérologie, Mougins
  - Hôpital Privé du Confluent SAS, Nantes
  - Hôpital Américain de Paris, Neuilly-sur-Seine
  - Hôpital Pierre Bérégovoy, Nevers
  - Centre Antoine Lacassagne, Nice
  - Centre Oncogard, Nîmes
  - CHU Carémeau, Nîmes
  - Hôpital de la Source, Orléans
  - Hôpital Privé des Peupliers, Paris
  - Hôpital Saint Antoine, Paris
  - HEGP, Paris
  - Hôpital Cochin, Paris
  - Hôpital Saint Louis, Paris
  - Institut Montsouris, Paris
  - Pitié Salpêtière, Paris
  - Centre Hospitalier, Pau
  - Hôpital Haut Leveque, Pessac
  - Polyclinique Francheville, Périgueux
  - CHU Lyon Sud, Pierre-Bénite
  - Centre CARIO - HCPA, Plérin
  - Hôpital de la Milétrie, Poitiers
  - CH Annecy Genevois, Pringy
  - CHU Robert Debré, Reims
  - CHU de Pontchaillou, Rennes
  - Centre Eugène Marquis, Rennes
  - CH, Rodez
  - Hôpital Drome Nord, Romans-sur-Isère
  - CHU Charles Nicolle, Rouen
  - Clinique Mathilde, Rouen
  - Institut Curie, Saint-Cloud
  - Hôpital Privé Saint Grégoire, Saint-Grégoire
  - ICO - Site René Gauducheau, Saint-Herblain
  - Polyclinique Côte Basque Sud, Saint-Jean-de-Luz
  - Hôpital d'Instruction des Armées Begin, Saint-Mandé
  - CH Région Saint Omer, Saint-Omer
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Polyclinique Saint Claude, Saint-Quentin
  - CH, Saint-Quentin
  - CH Saintonge, Saintes
  - CH Morlevat, Semur-en-Auxois
  - CH, Senlis
  - Centre Hospitalier, Sens
  - Centre Hospitalier de Saint-Malo, St-Malo
  - Clinique Sainte Anne, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Hôpitaux du Leman, Thonon-les-Bains
  - Hôpital Sainte Musse, Toulon
  - Clinique Saint Jean du Languedoc, Toulouse
  - Hôpitaux Trousseau, Tours
  - Centre Hospitalier, Valenciennes
  - CHU de Nancy-Bradois, Vandœuvre-lès-Nancy
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Paul Brousse, Villejuif
  - Centre Hospitalier, Villeneuve-Saint-Georges

REFERENCES:
- [Background] Aparicio T, Francois E, Cristol-Dalstein L, Carola E, Maillard E, Paillaud E, Retornaz F, Faroux R, Andre T, Bedenne L, Seitz JF. PRODIGE 34-FFCD 1402-ADAGE: Adjuvant chemotherapy in elderly patients with resected stage III colon cancer: A randomized phase 3 trial. Dig Liver Dis. 2016 Feb;48(2):206-7. doi: 10.1016/j.dld.2015.11.023. Epub 2015 Dec 2. No abstract available. PMID 26748426